CLINICAL TRIAL: NCT03079505
Title: Dasatinib Versus Nilotinib as Upfront Therapy for Treatment Naïve Chronic Myeloid Leukemia Chronic Phase
Brief Title: Dasatinib Versus Nilotinib for Treatment Naïve Chronic Myeloid Leukemia
Acronym: DANIN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Protocol Deviation
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17095/17
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-11

CONDITIONS: Chronic Myeloid Leukemia - Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dasatinib (Active Comparator): Dasatinib 100mg, once daily (QD), will be given to 25 patients, orally
  Interventions: Drug: Nilotinib 150mg oral capsule [Tasigna]
- Nilotinib (Experimental): Nilotinib 300mg, twice daily (BID), will be given to 25 patients, orally
  Interventions: Drug: Dasatinib 100 MG [Sprycel]

INTERVENTIONS:
Drug: Dasatinib 100 MG [Sprycel] — Dasatinib (Sprycel) 100 milligram, once-daily (QD) will be given to 25 patients orally
  Other Names: Sprycel
  Arms: Nilotinib
Drug: Nilotinib 150mg oral capsule [Tasigna] — Nilotinib (Tasigna) 300 milligram, twice-daily (BID) will be given to 25 patients orally
  Other Names: Tasigna
  Arms: Dasatinib

SUMMARY:
DANIN study is a randomized, phase 3 clinical trial comparing 'head to head' Nilotinib versus Dasatinib as upfront therapy for patient with chronic myeloid leukemia. The efficacy of both drugs will be tested by measuring BCR/ABL (BCR-ABL = fusion gene from BCR (breakpoint cluster region gene/BCR gene product) and ABL (Abelson proto-oncogene)) using European Leukemia net recommendations the study will be conducted in NCCCR (National Center for Cancer Care & Research) sample size calculations detailed in the statistic part the clinical hematologist will recruit the patients this will include consenting process inclusion and exclusion criteria the molecular pathologist will do the molecular testing the clinical research coordinator and fellows will do the CRF (Case Report Form) as well as quality of life questionnaire and applying the protocol for evaluation of cardiac evaluation Molecular monitoring of BCR-ABL1 transcripts to assess treatment response in CML (Chronic Myeloid Leukemia).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or over.
2. Patients must have all of the following:

   * be enrolled within 3 months of initial diagnosis of CML-CP (Chronic Phase) (date of initial diagnosis is the date of first cytogenetic analysis)
   * cytogenetic confirmation of the Philadelphia chromosome or variants of (9;22) translocations
   * patients may have secondary chromosomal abnormalities in addition to the Philadelphia chromosome.
   * < 15% blasts in peripheral blood and bone marrow;
   * < 30% blasts plus promyelocytes in peripheral blood and bone marrow;
   * < 20% basophils in peripheral blood,
   * 100 x 109/L platelets or greater
   * no evidence of extramedullary leukaemic involvement, with the exception of the hepatosplenomegaly.
3. Written voluntary informed consent.

Exclusion Criteria:

1 - Patients with Ph-negative, BCR-ABL-positive, disease are NOT eligible for the study.

2. Any prior treatment for CML with: any tyrosine kinase inhibitor (eg imatinib, dasatinib); busulphan; interferon-alpha; homoharringtonine; cytosine arabinoside; any other investigational agents (hydroxycarbamide and anagrelide are the only drugs permitted). Patients will be ineligible for the study if they have received any prior therapy with interferon-alpha or imatinib. No exceptions.

3. Patients who received prior chemotherapy, including regimens used in peripheral blood progenitor cells (PBPCs) mobilisation for haematopoietic progenitor-cell transplantation. (It is allowable to collect unmobilised PBPCs at diagnosis.) 4. Patient who have had any form of prior haemopoietic stem cell transplant, either autograft or allograft.

5. Patients with an ECOG (Eastern Cooperative Oncology Group) Performance Status Score of 2 or less.

6. Patients with serum bilirubin, AST (aspartate aminotransferase), ALT (alanine aminotransferase), or creatinine concentrations > 2.0 x the institutional upper limit of the normal range (IULN).

7. Patients with International normalized ratio (INR) or partial thromboplastin time (PTT) > 1.5 x IULN, with the exception of patients on treatment with oral anticoagulants.

8. Patients with uncontrolled medical disease such as diabetes mellitus, thyroid dysfunction, neuropsychiatric disorders, infection, angina, or Grade 3/4 cardiac problems as defined by the New York Heart Association Criteria.

9. Patients with known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required.

10. Patients who have undergone major surgery within 4 weeks of Study Day 1, or who have not recovered from prior major surgery.

11. Patients who are:

* pregnant,
* breast feeding,
* of childbearing potential without a negative pregnancy test prior to Study Day 1, and
* male or female of childbearing potential unwilling to use barrier contraceptive precautions throughout the trial (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).

  12. Patients with a history of another malignancy either currently or within the past five years, with the exception of basal cell skin carcinoma or cervical carcinoma in situ.

  13. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-09-23 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with a Molecular Response Rate (MMR) at 12 Months from the baseline | 12 Months
  Rate of MMR is defined as <= 0.1% BCR-ABL/ABL ratio by international scale (IS), measured by real-time quantitative polymerase chain reaction (RQ-PCR) which corresponds to a ≥ 3 log reduction of BCR-ABL transcript from standardized baseline. BCR-ABL = fusion gene from BCR (breakpoint cluster region gene/BCR gene product) and ABL (Abelson proto-oncogene)

SECONDARY OUTCOMES:
Number of patients with a Durable Molecular Response Rate (MMR) from the baseline | 12 months to 5 years
  Rate of MMR is defined as <= 0.1% BCR-ABL/ABL ratio by international scale (IS), measured by real-time quantitative polymerase chain reaction (RQ-PCR) which corresponds to a ≥ 3 log reduction of BCR-ABL transcript from standardized baseline. BCR-ABL = fusion gene from BCR (breakpoint cluster region gene/BCR gene product) and ABL (Abelson proto-oncogene) Number of patients with a maintained MMR for 5 years
Number of patients with a Reduction in BCR-ABL Transcript Levels in both arms from the baseline | 5 years
  BCR-ABL ≤ 10% at 3 months BCR-ABL < 1% at 6 months BCR-ABL ≤ 0.1% at 12 months
  then MMR or better
  BCR-ABL = fusion gene from BCR (breakpoint cluster region gene/BCR gene product) and ABL (Abelson proto-oncogene)
Number of patients with a Complete Cytogenetic Response (CCyR) in both arms from the baseline | 5 years
  Cytogenetic response (CyR) is based on the prevalence of Philadelphia positive (Ph+) cells in metaphase from bone marrow (BM) sample. (Ideally, 25 metaphases but at least 20 metaphases from a BM sample were evaluated). Complete Cytogenetic Response (CCyR)=0% Ph+ cells in metaphase in BM. A cCCyR=those in which all measurements up to at least 28 days after the initial response show an equivalent or better CCyR (Complete Cytogenetic Response).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Yassin, Principal Investigator — Hamad Medical Corporation
Locations (1):
- National Center for Cancer Care & Research (NCCCR), Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldman JM, Melo JV. Targeting the BCR-ABL tyrosine kinase in chronic myeloid leukemia. N Engl J Med. 2001 Apr 5;344(14):1084-6. doi: 10.1056/NEJM200104053441409. No abstract available. PMID 11287980
- [Background] Hehlmann R, Saussele S. Treatment of chronic myeloid leukemia in blast crisis. Haematologica. 2008 Dec;93(12):1765-9. doi: 10.3324/haematol.2008.001214. No abstract available. PMID 19050065
- [Background] Druker BJ, Guilhot F, O'Brien SG, Gathmann I, Kantarjian H, Gattermann N, Deininger MW, Silver RT, Goldman JM, Stone RM, Cervantes F, Hochhaus A, Powell BL, Gabrilove JL, Rousselot P, Reiffers J, Cornelissen JJ, Hughes T, Agis H, Fischer T, Verhoef G, Shepherd J, Saglio G, Gratwohl A, Nielsen JL, Radich JP, Simonsson B, Taylor K, Baccarani M, So C, Letvak L, Larson RA; IRIS Investigators. Five-year follow-up of patients receiving imatinib for chronic myeloid leukemia. N Engl J Med. 2006 Dec 7;355(23):2408-17. doi: 10.1056/NEJMoa062867. PMID 17151364
- [Background] Deininger M, O'Brien SG, Guilhot F, et al. International randomized study of interferon vs STI571 (IRIS) 8-year follow up: sustained survival and low risk for progression or events in patients with newly diagnosed chronic myeloid leukemia in chronic phase treated with imatinib [abstract]. Blood (ASH Annual Meeting Abstracts) 2009;114(22). Abstract 1126.
- [Background] de Lavallade H, Apperley JF, Khorashad JS, Milojkovic D, Reid AG, Bua M, Szydlo R, Olavarria E, Kaeda J, Goldman JM, Marin D. Imatinib for newly diagnosed patients with chronic myeloid leukemia: incidence of sustained responses in an intention-to-treat analysis. J Clin Oncol. 2008 Jul 10;26(20):3358-63. doi: 10.1200/JCO.2007.15.8154. Epub 2008 Jun 2. PMID 18519952
- [Background] O'Hare T, Walters DK, Stoffregen EP, Jia T, Manley PW, Mestan J, Cowan-Jacob SW, Lee FY, Heinrich MC, Deininger MW, Druker BJ. In vitro activity of Bcr-Abl inhibitors AMN107 and BMS-354825 against clinically relevant imatinib-resistant Abl kinase domain mutants. Cancer Res. 2005 Jun 1;65(11):4500-5. doi: 10.1158/0008-5472.CAN-05-0259. PMID 15930265
- [Background] Cortes JE, Kim DW, Pinilla-Ibarz J, le Coutre P, Paquette R, Chuah C, Nicolini FE, Apperley JF, Khoury HJ, Talpaz M, DiPersio J, DeAngelo DJ, Abruzzese E, Rea D, Baccarani M, Muller MC, Gambacorti-Passerini C, Wong S, Lustgarten S, Rivera VM, Clackson T, Turner CD, Haluska FG, Guilhot F, Deininger MW, Hochhaus A, Hughes T, Goldman JM, Shah NP, Kantarjian H; PACE Investigators. A phase 2 trial of ponatinib in Philadelphia chromosome-positive leukemias. N Engl J Med. 2013 Nov 7;369(19):1783-96. doi: 10.1056/NEJMoa1306494. Epub 2013 Nov 1. PMID 24180494
- [Background] Cortes JE, Jones D, O'Brien S, Jabbour E, Ravandi F, Koller C, Borthakur G, Walker B, Zhao W, Shan J, Kantarjian H. Results of dasatinib therapy in patients with early chronic-phase chronic myeloid leukemia. J Clin Oncol. 2010 Jan 20;28(3):398-404. doi: 10.1200/JCO.2009.25.4920. Epub 2009 Dec 14. PMID 20008620
- [Background] Kantarjian H, Shah NP, Hochhaus A, Cortes J, Shah S, Ayala M, Moiraghi B, Shen Z, Mayer J, Pasquini R, Nakamae H, Huguet F, Boque C, Chuah C, Bleickardt E, Bradley-Garelik MB, Zhu C, Szatrowski T, Shapiro D, Baccarani M. Dasatinib versus imatinib in newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2010 Jun 17;362(24):2260-70. doi: 10.1056/NEJMoa1002315. Epub 2010 Jun 5. PMID 20525995